CLINICAL TRIAL: NCT02535364
Title: A Phase 2, Single-arm, Multicenter Trial to Determine the Efficacy and Safety of JCAR015 in Adult Subjects With Relapsed or Refractory B-Cell Acute Lymphoblastic Leukemia
Brief Title: Study Evaluating the Efficacy and Safety of JCAR015 in Adult B-cell Acute Lymphoblastic Leukemia (B-ALL)
Acronym: ROCKET
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Safety reasons
Sponsor: Juno Therapeutics, a Subsidiary of Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 015001
Record Dates: First submitted 2015-08-24; First posted 2015-08-28 (Estimated); Results first posted 2018-07-19 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: acute lymphoblastic leukemia; ALL; chimeric antigen receptor; CAR; CAR T cells; JCAR015; autologous T cell therapy; cell therapy
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- JCAR015 (CD19-targeted CAR T cells) (Experimental): JCAR015 was administered as two intravenous (IV) infusions separated by 14 to 28 days.
  Interventions: Biological: JCAR015 (CD19-targeted CAR T cells)

INTERVENTIONS:
Biological: JCAR015 (CD19-targeted CAR T cells) — Part A: Following leukapheresis and concurrent with generation of JCAR015, participants received, at the Investigator's discretion, cytoreductive chemotherapy based on the Investigator's choice of regimens and/or supportive care.
  Part B: Participants who were eligible for treatment in Part B received two IV doses of JCAR015 CAR T cells separated by 14 to 28 days. JCAR015 infusion was preceded by lymphodepleting chemotherapy with cyclophosphamide alone or cyclophosphamide + fludarabine.

SUMMARY:
This single-arm, multicenter Phase 2 trial will treat adult patients who have relapsed or refractory B-ALL with an infusion of the patient's own T cells that have been genetically modified to express a chimeric antigen receptor (CAR) that will bind to leukemia cells that express the CD19 protein on the cell surface. The study will determine if these modified T cells (called JCAR015) help the body's immune system eliminate leukemia cells. The trial will also study the safety of treatment with JCAR015, how long JCAR015 cells stay in the patient's body, the extent to which JCAR015 eliminates minimal residual disease, and the impact of this treatment on survival.

DETAILED DESCRIPTION:
This is a single-arm, multicenter Phase 2 study to determine the efficacy and safety of JCAR015 in adult patients with relapsed or refractory B-ALL. The study will have the following sequential phases: Part A (screening, leukapheresis, cell product preparation, and cytoreductive chemotherapy) and Part B (treatment and follow-up). The follow-up period for each participant is approximately 12 months after the final JCAR015 infusion. The total duration of the study is expected to be approximately 3 years. Long-term follow-up for survival, toxicity, and viral vector safety will continue under a separate long-term follow-up protocol per health regulatory authority guidelines, currently up to 15 years after the last JCAR015 infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of consent
2. Relapsed or refractory B-ALL, defined as:

   * First or greater bone marrow relapse from CR, or
   * Any bone marrow relapse after allogeneic hematopoietic stem cell transplant (HSCT); subjects must be at least 100 days from HSCT at the time of screening and off immunosuppressant medication for at least 1 month at the time of screening, and have no active graft-vs-host disease (GVHD), or
   * Refractory B-ALL, defined by not having achieved a CR or CRi after two attempts at remission induction using standard regimens, or
   * Ph+ B-ALL if subjects are intolerant to or ineligible for tyrosine kinase inhibitor (TKI) therapy, or have progressed after at least one line of TKI therapy
3. Morphological evidence of disease in bone marrow (at least 5% blasts)
4. Evidence of CD19 expression
5. Eastern Cooperative Oncology Group (ECOG) performance status between 0 and 2 at the time of screening
6. Adequate pulmonary, renal, hepatic, and cardiac function
7. Adequate central or peripheral vascular access for leukapheresis procedure

Exclusion Criteria:

1. Isolated extramedullary disease relapse
2. Concomitant genetic syndrome or other known bone marrow failure syndrome
3. Burkitt's lymphoma/leukemia or chronic myelogenous leukemia lymphoid blast crisis (p210 BCR-ABL+)
4. Prior malignancy, unless treated with curative intent and with no evidence of active disease present for > 5 years before screening
5. Prior treatment with any gene therapy product
6. Active hepatitis B, active hepatitis C, or any human immunodeficiency virus (HIV) infection at the time of screening
7. Systemic fungal, bacterial, viral, or other infection that is not controlled, at the time of screening
8. Presence of Grade II-IV (Glucksberg) or B-D (IBMTR) acute or extensive chronic GVHD at the time of screening
9. Active central nervous system (CNS) involvement by malignancy (defined as CNS-3 per National Comprehensive Cancer Network [NCCN] guidelines)
10. History of any one of the following cardiovascular conditions within the past 6 months: Class III or IV heart failure as defined by the New York Heart Association (NYHA), cardiac angioplasty or stenting, myocardial infarction, unstable angina, or other clinically significant cardiac disease
11. History or presence of clinically relevant CNS pathology such as epilepsy, generalized seizure disorder, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis
12. Participation in an investigational research study using an investigational agent within 30 days of screening
13. History of treatment with a murine-derived biological product other than blinatumomab unless subject has been shown to be negative for human-anti-mouse-antibodies (HAMA) prior to or during screening
14. Pregnant or nursing women
15. Use of prohibited medications:

    1. Steroids: Therapeutic doses of corticosteroids are prohibited within 7 days prior to leukapheresis.
    2. Allogeneic cellular therapy: Donor lymphocyte infusions (DLI) are prohibited within 4 weeks prior to leukapheresis
    3. GVHD therapies: Any drug used for GVHD within 4 weeks prior to leukapheresis
    4. Chemotherapies: Salvage chemotherapy must be stopped at least 1 week prior to leukapheresis
16. Treatment with alemtuzumab within 6 months prior to leukapheresis, or treatment with clofarabine or cladribine within 3 months prior to leukapheresis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2015-08-21 (Actual); Primary Completion 2017-04-24 (Actual); Study Completion 2017-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaus Trede, MD, PhD, Study Director — Juno Therapeutics, Inc., a Bristol-Myers Squibb Company
Locations (18):
- United States (18):
  - University of Alabama Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - City of Hope, Duarte, California
  - University of California, San Francisco, California
  - University of Colorado Denver -- Anschutz Medical Campus, Aurora, Colorado
  - Sylvester Comprehensive Cancer Center/UMHC, Miami, Florida
  - The Blood and Marrow Transplant Program at Northside Hospital, Atlanta, Georgia
  - Northwestern University Robert H Lurie Comprehensive Cancer Center, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Sidney Kimmel Comprehensive Cancer Center @ Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Background] Davila ML, Riviere I, Wang X, Bartido S, Park J, Curran K, Chung SS, Stefanski J, Borquez-Ojeda O, Olszewska M, Qu J, Wasielewska T, He Q, Fink M, Shinglot H, Youssif M, Satter M, Wang Y, Hosey J, Quintanilla H, Halton E, Bernal Y, Bouhassira DC, Arcila ME, Gonen M, Roboz GJ, Maslak P, Douer D, Frattini MG, Giralt S, Sadelain M, Brentjens R. Efficacy and toxicity management of 19-28z CAR T cell therapy in B cell acute lymphoblastic leukemia. Sci Transl Med. 2014 Feb 19;6(224):224ra25. doi: 10.1126/scitranslmed.3008226. PMID 24553386
- [Background] Sadelain M, Brentjens R, Riviere I. The basic principles of chimeric antigen receptor design. Cancer Discov. 2013 Apr;3(4):388-98. doi: 10.1158/2159-8290.CD-12-0548. Epub 2013 Apr 2. PMID 23550147
- [Background] Brentjens RJ, Davila ML, Riviere I, Park J, Wang X, Cowell LG, Bartido S, Stefanski J, Taylor C, Olszewska M, Borquez-Ojeda O, Qu J, Wasielewska T, He Q, Bernal Y, Rijo IV, Hedvat C, Kobos R, Curran K, Steinherz P, Jurcic J, Rosenblat T, Maslak P, Frattini M, Sadelain M. CD19-targeted T cells rapidly induce molecular remissions in adults with chemotherapy-refractory acute lymphoblastic leukemia. Sci Transl Med. 2013 Mar 20;5(177):177ra38. doi: 10.1126/scitranslmed.3005930. PMID 23515080
- [Background] Brentjens RJ, Riviere I, Park JH, Davila ML, Wang X, Stefanski J, Taylor C, Yeh R, Bartido S, Borquez-Ojeda O, Olszewska M, Bernal Y, Pegram H, Przybylowski M, Hollyman D, Usachenko Y, Pirraglia D, Hosey J, Santos E, Halton E, Maslak P, Scheinberg D, Jurcic J, Heaney M, Heller G, Frattini M, Sadelain M. Safety and persistence of adoptively transferred autologous CD19-targeted T cells in patients with relapsed or chemotherapy refractory B-cell leukemias. Blood. 2011 Nov 3;118(18):4817-28. doi: 10.1182/blood-2011-04-348540. Epub 2011 Aug 17. PMID 21849486

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 82 participants were enrolled at 15 study centers within the United States.
Pre-assignment Details: Participants were adults with relapsed or refractory CD19-positive B-cell acute lymphoblastic leukemia (ALL).
Groups:
- JCAR015: Participants received up to two intravenous (IV) infusions of JCAR015 separated by 14 to 28 days. In Part A, participants received at the Investigator's discretion, cytoreductive chemotherapy based on the Investigator's choice and/or supportive care. In Part B, eligible participants received two IV doses of JCAR015 CAR T cells. JCAR015 infusion was preceded by lymphodepleting chemotherapy with cyclophosphamide alone or cyclophosphamide + fludarabine.
Period: Part A Screening Through Leukapheresis
Arm/Group | JCAR015
Started | 82
Completed | 57
Not Completed | 25
Not completed — Failure to meet criteria for Part A | 22
Not completed — Study placed on clinical hold by FDA | 2
Not completed — Disease progression | 1
Period: Part B Screening
Arm/Group | JCAR015
Started | 57
Completed | 40
Not Completed | 17
Not completed — Study placed on clinical hold by FDA | 7
Not completed — Unable to manufacture JCAR015 | 3
Not completed — Death | 2
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1
Not completed — Change in diagnosis, no longer eligible | 2
Period: Study Treatment
Arm/Group | JCAR015
Started | 40
Completed | 38
Not Completed | 2
Not completed — Death | 1
Not completed — Study placed on clinical hold by FDA | 1
Period: 12-Month Follow-up Period
Arm/Group | JCAR015
Started | 38
Completed | 3
Not Completed | 35
Not completed — Disease progression | 22
Not completed — Death | 5
Not completed — Underwent stem cell transplant | 5
Not completed — Subject received alternative therapy | 2
Not completed — Subject transferred to hospice | 1

BASELINE CHARACTERISTICS:
Population: Total number of subjects who received at least one infusion of JCAR015
Groups:
- JCAR015: Participants received up to two IV infusions of JCAR015 separated by 14 to 28 days.
Arm/Group | JCAR015
Number analyzed (Participants) | 38
Age, Continuous [Median (Full Range); unit: years] | 39 [19 to 69]
Age, Customized [Count of Participants; unit: Participants]
  39 or younger | 19
  40 to 64 | 15
  65 or older | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 35
  More than one race | 0
  Unknown or Not Reported | 0
Time Since Diagnosis [Median (Full Range); unit: years] | 1.8 [1 to 22]
Number of Prior Lines of Therapy [Median (Full Range); unit: lines of therapy] | 2 [1 to 7]
Most Recent Prior Regimen [Count of Participants; unit: Participants]
  Blinatumomab monotherapy | 11
  Investigational agent | 1
  Marqibo | 2
  Multi-agent chemotherapy | 15
  Tyrosine kinase inhibitor + chemotherapy | 2
  Tyrosine kinase inhibitor alone | 1
  Other | 6
Response to Most Recent Prior Regimen [Count of Participants; unit: Participants]
  Remission | 8
  No response | 27
  Not applicable | 2
  Missing | 1
Prior Stem Cell Transplant [Count of Participants; unit: Participants]
  Received prior stem cell transplant | 14
  Did not receive prior stem cell transplant | 24
Eastern Cooperative Oncology Group (ECOG) Score [Count of Participants; unit: Participants] — 0 = Fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, eg, light house work, office work; 2 = Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about > 50% of waking hours; 3 = Capable of only limited self-care, confined to bed or chair > 50% of waking hours; 4 = Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair
  From Oken MM, et al. Am J Clin Oncol 1982;5(6):649-655.
  Participants
    0 | 3
    1 | 29
    2 | 5
    3 | 1
Philadelphia Chromosome Status [Count of Participants; unit: Participants] — The Philadelphia (Ph) chromosome is an abnormally short chromosome 22 that results from translocation between the BCR gene on chromosome 22 with the ABL gene on chromosome 9. The resulting BCR-ABL gene encodes a fusion protein with uncontrolled tyrosine kinase activity and has been linked to chronic myeloid leukemia and one form of ALL.
  Participants
    Philadelphia chromosome negative | 34
    Philadelphia chromosome positive | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Remission (CR) or Complete Remission With Incomplete Hematopoietic Recovery (CRi), as Determined by an Independent Review Committee (IRC)
Description: Overall remission rate (ORR) is defined as the percentage of participants with CR or CRi based on IRC assessment. For CR, all of the following must be met: (1) in bone marrow, trilineage hematopoiesis and < 5% blasts; (2) in peripheral blood, neutrophils > 1,000/µL, platelets > 100,000/µL, and circulating blasts < 1%; (3) no clinical evidence of extramedullary disease by physical examination and no symptoms suggestive of CNS involvement (if additional assessments such as CSF assessment by lumbar puncture or Ommaya reservoir tap, CNS imaging, or biopsy are performed, results must show no evidence of disease); (4) no platelet and/or neutrophil transfusions ≤ 7 days before the date of peripheral blood sampling, and (5) no clinical evidence of recurrence for 4 weeks. For CRi, all criteria for CR are met except that one or more of the following exists in the peripheral blood: neutrophils ≤ 1,000/µL, platelets ≤ 100,000/µL, or platelet transfusions ≤ 7 days before blood sampling.
Time Frame: Day 1 (first JCAR015 infusion) up to 12 months after the last JCAR015 infusion
Population: The analysis population includes participants with morphological disease at the time of the first JCAR015 infusion who received lymphodepleting chemotherapy with cyclophosphamide alone and at least one JCAR015 infusion, and who were evaluable for response (excludes 2 subjects with Grade 5 brain edema who died within 8 days after JCAR015 infusion).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JCAR015
Number analyzed (Participants) | 22
percentage of participants | 45.5 [24.4 to 67.8]

2. Secondary Outcome: Percentage of Participants With CR or CRi, as Determined by an IRC
Description: ORR is defined as the percentage of participants with CR or CRi based on IRC assessment (refer to criteria in Outcome Measure #1)
Time Frame: Day 1 (first JCAR015 infusion) up to 12 months after the last JCAR015 infusion
Population: The analysis population includes participants with morphologic disease who received lymphodepleting chemotherapy with cyclophosphamide alone or cyclophosphamide + fludarabine and at least one JCAR015 infusion, and who were evaluable for response (excludes 5 subjects with Grade 5 brain edema who died within 8 days after JCAR015 infusion).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JCAR015
Number analyzed (Participants) | 27
percentage of participants | 55.6 [35.3 to 74.5]

3. Secondary Outcome: Percentage of Participants Who Achieved a CR or CRi, as Determined by an IRC
Description: Best overall response (BOR) is defined as the best disease response recorded from the time of the last JCAR015 infusion until the start of another anticancer therapy (refer to Outcome Measure #1 for criteria for CR and CRi).
Time Frame: Day 1 (first JCAR015 infusion) up to 12 months after the last JCAR015 infusion
Population: The analysis population includes all participants with morphological disease at the time of the first JCAR015 infusion who received lymphodepleting chemotherapy with cyclophosphamide alone and at least one infusion of JCAR015.
Measure: Number; unit: percentage of participants
Arm/Group | JCAR015
Number analyzed (Participants) | 24
percentage of participants
  CR | 8.3
  CRi | 33.3

4. Secondary Outcome: Percentage of Participants Who Achieved a CR or CRi, as Determined by an IRC
Description: BOR is defined as the best disease response recorded from the time of the last JCAR015 infusion until the start of another anticancer therapy (refer to Outcome Measure #1 for criteria for CR and CRi).
Time Frame: Day 1 (first JCAR015 infusion) up to 12 months after the last JCAR015 infusion
Population: The analysis population includes all participants with morphologic disease at the time of JCAR015 infusion who received lymphodepleting chemotherapy with cyclophosphamide alone or cyclophosphamide + fludarabine and at least one infusion of JCAR015.
Measure: Number; unit: percentage of participants
Arm/Group | JCAR015
Number analyzed (Participants) | 32
percentage of participants
  CR | 12.5
  CRi | 34.3

5. Secondary Outcome: Percentage of Participants Who Achieved a Minimal Residual Disease (MRD)-Negative CR or CRi
Description: Percentage of participants who achieved a CR or CRi, as determined by an IRC, with no evidence of MRD in the bone marrow (refer to Outcome Measure #1 for criteria for CR and CRi). MRD-negative is defined as undetectable leukemic cells in the bone marrow as determined by a polymerase chain reaction (PCR)-based assay.
Time Frame: Day 1 (first JCAR015 infusion) up to 12 months after the last JCAR015 infusion
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | JCAR015
Number analyzed (Participants) | 24
percentage of participants
  MRD-negative CR/CRi | 41.7
  MRD-positive CR/CRi | 0
  MRD-negative CR/CRi unconfirmed | 12.6
  MRD-positive CR/CRi unconfirmed | 4.2

6. Secondary Outcome: Percentage of Participants Who Achieved a MRD-Negative CR or CRi
Description: Percentage of participants who achieved a CR or CRi, as determined by an IRC, with no evidence of MRD in the bone marrow (refer to Outcome Measure #1 for criteria for CR and CRi). MRD-negative is defined as undetectable leukemic cells in the bone marrow as determined by a PCR-based assay.
Time Frame: Day 1 (first JCAR015 infusion) up to 12 months after the last JCAR015 infusion
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | JCAR015
Number analyzed (Participants) | 32
percentage of participants
  MRD-negative CR/CRi | 46.9
  MRD-positive CR/CRi | 0
  MRD-negative CR/CRi unconfirmed | 9.4
  MRD-positive CR/CRi unconfirmed | 3.1

7. Secondary Outcome: Relapse-Free Survival (RFS), as Determined by an IRC
Description: RFS is defined as the interval from the first documentation of CR or CRi (refer to Outcome Measure #1) to the earlier date of relapse or death due to any cause. Participants who proceeded to hematopoietic stem cell transplant (HSCT) after JCAR015 infusion were censored at the time of HSCT.
Time Frame: Day 1 (first JCAR015 infusion) up to 12 months after the last JCAR015 infusion
Population: The analysis population includes participants with morphological disease at the time of the first JCAR015 infusion who received lymphodepleting chemotherapy with cyclophosphamide alone and at least one infusion of JCAR015, and who achieved a CR or CRi after JCAR015 infusion.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | JCAR015
Number analyzed (Participants) | 10
months | 6.3 [1.9 to NA] — The upper limit of the 95% confidence interval was not reached.

8. Secondary Outcome: RFS, as Determined by an IRC
Description: RFS is defined as the interval from the first documentation of CR or CRi (refer to Outcome Measure #1) to the earlier date of relapse or death due to any cause. Participants who proceeded to HSCT after JCAR015 infusion were censored at the time of HSCT.
Time Frame: Day 1 (first JCAR015 infusion) up to 12 months after the last JCAR015 infusion
Population: The analysis population includes participants with morphologic disease at the time of JCAR015 infusion who received lymphodepleting chemotherapy with cyclophosphamide alone or cyclophosphamide + fludarabine and at least one infusion of JCAR015, and who achieved a CR or CRi after JCAR015 infusion.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | JCAR015
Number analyzed (Participants) | 15
months | 4.4 [2.1 to 9.4]

9. Secondary Outcome: Event-Free Survival (EFS)
Description: EFS is defined as the time from the date of the first JCAR015 infusion to the earliest of the following events: death from any cause, relapse, or treatment failure (defined as no response and subsequent discontinuation from the study for adverse event, lack of efficacy or progressive disease, or new anticancer therapy). Participants who proceeded to HSCT after JCAR015 infusion were censored at the time of HSCT.
Time Frame: Day 1 (first JCAR015 infusion) up to 12 months after the last JCAR015 infusion
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | JCAR015
Number analyzed (Participants) | 24
months | 0.03 [0.03 to 3.8]

10. Secondary Outcome: EFS
Description: as for outcome 9
Time Frame: Day 1 (first JCAR015 infusion) up to 12 months after the last JCAR015 infusion
Population: The analysis population includes all participants who received lymphodepleting chemotherapy with cyclophosphamide alone or cyclophosphamide + fludarabine and at least one infusion of JCAR015.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | JCAR015
Number analyzed (Participants) | 38
months | 2.7 [0.03 to 4.2]

11. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the interval from the date of the first JCAR015 infusion to the date of death due to any reason.
Time Frame: Day 1 (first JCAR015 infusion) up to 12 months after the last JCAR015 infusion
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | JCAR015
Number analyzed (Participants) | 24
months | 7.33 [5.16 to 12.68]

12. Secondary Outcome: OS
Description: OS is defined as the interval from the date of the first JCAR015 infusion to the date of death due to any reason.
Time Frame: Day 1 (first JCAR015 infusion) up to 12 months after the last JCAR015 infusion
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | JCAR015
Number analyzed (Participants) | 38
months | 8.15 [5.32 to 12.68]

13. Secondary Outcome: Duration of Remission (DOR) as Determined by an IRC
Description: DOR is defined as the interval from the first documentation of CR or CRi to the earlier date of relapse or death due to ALL.
Time Frame: Day 1 (first JCAR015 infusion) up to 12 months after the last JCAR015 infusion
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | JCAR015
Number analyzed (Participants) | 15
months | 4.4 [2.1 to 9.4]

14. Secondary Outcome: Percentage of Participants Who Achieved a CR or CRi, as Determined by an IRC, at Month 6 After the Final JCAR015 Infusion
Description: ORR at Month 6 is defined as the percentage of participants who achieved a CR or CRi at Month 6 after the final JCAR015 infusion without HSCT during the time period between the final JCAR015 infusion and the Month 6 response assessment (refer to Outcome Measure #1 for criteria for CR and CRi).
Time Frame: Day 1 (first JCAR015 infusion) up to 6 months after the last JCAR015 infusion
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | JCAR015
Number analyzed (Participants) | 32
percentage of participants
  Maintained CR at Month 6 | 11.1
  Maintained CRi at Month 6 | 3.7

15. Secondary Outcome: Percentage of Participants Who Achieved a Morphologic Remission Within 6 Months After the Final JCAR015 Infusion and Then Proceeded to HSCT
Description: Percentage of participants who achieved a morphologic remission within 6 months after the final JCAR015 infusion and then proceeded to HSCT prior to 12 months after the final JCAR015 infusion
Time Frame: Day 1 (first JCAR015 infusion) up to 12 months after the last JCAR015 infusion
Population: The analysis population includes participants with morphologic disease at the time of JCAR015 infusion who received lymphodepleting chemotherapy with cyclophosphamide alone or cyclophosphamide + fludarabine and at least one infusion of JCAR015, and who were evaluable for response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JCAR015
Number analyzed (Participants) | 27
percentage of participants | 11.1 [2.4 to 29.2]

16. Secondary Outcome: Maximum Concentration of JCAR015 (Cmax) in the Peripheral Blood by Quantitative Polymerase Chain Reaction (qPCR)
Description: Cmax is defined as the highest measured number of copies of JCAR015 transgene per microgram of genomic DNA in peripheral blood cells as assessed by qPCR.
Time Frame: Pre-dose Day 1 of each JCAR015 infusion; Day 4, Day 7, Day 14, Day 21, and Day 28 after the first JCAR015 infusion until receipt of the second infusion; and Day 4, Day 7, Day 14, Day 21, and Day 28 after the second JCAR015 infusion (if applicable)
Population: The analysis population includes all participants who received at least one infusion of JCAR015.
Measure: Median (Full Range); unit: vector copy number/microgram
Arm/Group | JCAR015
Number analyzed (Participants) | 38
vector copy number/microgram | 69246 [32 to 408583]

17. Secondary Outcome: Maximum Concentration of JCAR015 (Cmax) in the Peripheral Blood by Flow Cytometry
Description: Cmax is defined as the highest measured concentration of JCAR015 CAR T cells per microliter of peripheral blood as measured by flow cytometry.
Time Frame: as for outcome 16
Population: The analysis population includes all participants who received at least one infusion of JCAR015.
Measure: Median (Full Range); unit: cells/microliter
Arm/Group | JCAR015
Number analyzed (Participants) | 38
cells/microliter | 8.1 [0 to 556]

18. Secondary Outcome: Time to Maximum Concentration of JCAR015 (Tmax) in the Peripheral Blood as Measured by qPCR
Description: Tmax is defined as the time after the JCAR015 infusion at which the maximum concentration (Cmax) as measured by qPCR is observed. If Cmax occurred after the second infusion, Tmax was calculated from the time of the second infusion.
Time Frame: as for outcome 16
Population: The analysis population includes all participants who received at least one infusion of JCAR015.
Measure: Median (Full Range); unit: days
Arm/Group | JCAR015
Number analyzed (Participants) | 38
days | 8 [4 to 18]

19. Secondary Outcome: Tmax in the Peripheral Blood as Measured by Flow Cytometry
Description: Tmax is defined as the time after the JCAR015 infusion at which the Cmax as measured by flow cytometry of the JCAR015 CAR is observed. If Cmax occurred after the second infusion, Tmax was calculated from the time of the second infusion.
Time Frame: as for outcome 16
Population: The analysis population includes all participants who received at least one infusion of JCAR015 and whose Cmax was >0.
Measure: Median (Full Range); unit: days
Arm/Group | JCAR015
Number analyzed (Participants) | 34
days | 10.5 [6 to 29]

20. Secondary Outcome: Area Under the Concentration-vs-Time Curve (AUC) for JCAR015 in the Peripheral Blood as Measured by qPCR
Description: AUC is defined as the area under the concentration-vs-time curve from Day 1 to Day 29 after the first JCAR015 infusion as measured by qPCR of the JCAR015 transgene. AUC calculation includes pharmacokinetic (PK) results up to the second JCAR015 infusion for subjects who received the second infusion prior to Day 29 after the first JCAR015 infusion.
Time Frame: Pre-dose Day 1 of the first JCAR015 infusion; Day 4, Day 7, Day 14, Day 21, and Day 28 after the first JCAR015 infusion until receipt of the second infusion
Population: The analysis population includes all participants who received at least one infusion of JCAR015.
Measure: Median (Full Range); unit: vector copy number*days/microgram
Arm/Group | JCAR015
Number analyzed (Participants) | 38
vector copy number*days/microgram | 556520 [96 to 4628485]

21. Secondary Outcome: AUC for JCAR015 in the Peripheral Blood as Measured by Flow Cytometry
Description: AUC is defined as the area under the concentration-vs-time curve from Day 1 to Day 29 after the first JCAR015 infusion as measured by flow cytometry of the JCAR015 CAR. AUC calculation includes PK results up to the second JCAR015 infusion for subjects who received the second infusion prior to Day 29 after the first JCAR015 infusion.
Time Frame: as for outcome 20
Population: The analysis population includes all participants who received at least one infusion of JCAR015.
Measure: Median (Full Range); unit: cells*days/microliter
Arm/Group | JCAR015
Number analyzed (Participants) | 38
cells*days/microliter | 60.6 [0 to 6806]

22. Secondary Outcome: Percentage of Participants Who Developed Anti-Therapeutic Antibodies Against JCAR015
Description: Percentage of participants who developed anti-therapeutic antibodies against JCAR015
Time Frame: Part B Screening; Day 14 after the first JCAR015 infusion; Pre-Dose Day 1 of the second JCAR015 infusion; Day 14 after the second JCAR015 infusion; and Day 28, Month 3, Month 6, and Month 12 after the last JCAR015 infusion
Population: The analysis population includes all enrolled subjects who underwent leukapheresis and had a sample that was evaluable for the assay.
Measure: Number; unit: percentage of participants
Arm/Group | JCAR015
Number analyzed (Participants) | 41
percentage of participants
  Day 28 after last infusion: number analyzed (Participants) | 21
  Day 28 after last infusion | 10
  Month 3: number analyzed (Participants) | 14
  Month 3 | 64
  Month 6: number analyzed (Participants) | 6
  Month 6 | 83
  Month 12: number analyzed (Participants) | 9
  Month 12 | 22

ADVERSE EVENTS:
Time Frame: From the time of the first JCAR015 infusion up to 12 months after the last JCAR015 infusion
Description: The summary tables include treatment-emergent adverse events, defined as adverse events that (1) occurred or worsened after the first JCAR015 infusion and up to 30 days after the final JCAR015 infusion or (2) led to JCAR015 discontinuation. Adverse events occurring after the initiation of another anticancer therapy were not considered as treatment-emergent adverse events.
Arm/Group | JCAR015
All-Cause Mortality (participants affected / at risk) | 24/38
Serious Adverse Events (participants affected / at risk) | 23/38
Other Adverse Events (participants affected / at risk) | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | JCAR015 (N=38)
Encephalopathy (Nervous system disorders) | 8
Cytokine release syndrome (Immune system disorders) | 8
Brain oedema (Nervous system disorders) | 5
Seizure (Nervous system disorders) | 2
Sepsis (Infections and infestations) | 2
Generalised tonic-clonic seizure (Nervous system disorders) | 1
Bacteraemia (Infections and infestations) | 1
Fungaemia (Infections and infestations) | 1
Neutropenic colitis (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Pyrexia (General disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | JCAR015 (N=38)
Cytokine release syndrome (Immune system disorders) | 29
Confusional state (Psychiatric disorders) | 18
Diarrhoea (Gastrointestinal disorders) | 17
Nausea (Gastrointestinal disorders) | 16
Aphasia (Nervous system disorders) | 15
Vomiting (Gastrointestinal disorders) | 15
Tremor (Nervous system disorders) | 12
Headache (Nervous system disorders) | 10
Hypokalaemia (Metabolism and nutrition disorders) | 10
Somnolence (Nervous system disorders) | 10
Anaemia (Blood and lymphatic system disorders) | 9
Fatigue (General disorders) | 9
Decreased appetite (Metabolism and nutrition disorders) | 8
Hypomagnesaemia (Metabolism and nutrition disorders) | 8
Insomnia (Psychiatric disorders) | 8
Lethargy (Nervous system disorders) | 8
Muscular weakness (Musculoskeletal and connective tissue disorders) | 8
Chills (General disorders) | 7
Neutrophil count decreased (Investigations) | 7
Oedema peripheral (General disorders) | 7
Platelet count decreased (Investigations) | 7
Seizure (Nervous system disorders) | 7
Agitation (Psychiatric disorders) | 6
Asthenia (General disorders) | 6
Delirium (Psychiatric disorders) | 6
Depressed level of consciousness (Nervous system disorders) | 6
Encephalopathy (Nervous system disorders) | 6
Febrile neutropenia (Blood and lymphatic system disorders) | 6
Hypertension (Vascular disorders) | 6
White blood cell count decreased (Investigations) | 6
Anxiety (Psychiatric disorders) | 5
Constipation (Gastrointestinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Pyrexia (General disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4
Blood bilirubin increased (Investigations) | 4
Dizziness (Nervous system disorders) | 4
Fall (Injury, poisoning and procedural complications) | 4
Gait disturbance (General disorders) | 4
Haematuria (Renal and urinary disorders) | 4
Mental status changes (Psychiatric disorders) | 4
Oedema (Respiratory, thoracic and mediastinal disorders) | 4
Peripheral sensory neuropathy (Nervous system disorders) | 4
Pneumonia (Infections and infestations) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 4
Staphylococcal infection (Infections and infestations) | 4
Abdominal distension (Gastrointestinal disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Candida infection (Infections and infestations) | 3
Depression (Psychiatric disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Fluid overload (Metabolism and nutrition disorders) | 3
Hallucination (Psychiatric disorders) | 3
Hypoaesthesia (Nervous system disorders) | 3
Hyponatraemia (Metabolism and nutrition disorders) | 3
Hypotension (Vascular disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Memory impairment (Nervous system disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 3
Night sweats (Skin and subcutaneous tissue disorders) | 3
Pain (General disorders) | 3
Photophobia (Eye disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Sinus bradycardia (Cardiac disorders) | 3
Urinary incontinence (Renal and urinary disorders) | 3
Urinary retention (Renal and urinary disorders) | 3
Abdominal discomfort (Gastrointestinal disorders) | 2
Abdominal pain lower (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 2
Alanine aminotransferase increased (Investigations) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2
Angina pectoris (Cardiac disorders) | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Ataxia (Nervous system disorders) | 2
Blood alkaline phosphatase increased (Investigations) | 2
Blood bicarbonate decreased (Investigations) | 2
Blood creatinine increased (Investigations) | 2
Blood fibrinogen decreased (Investigations) | 2
Bradycardia (Cardiac disorders) | 2
Catheter site pain (General disorders) | 2
Cellulitis (Infections and infestations) | 2
Chest discomfort (General disorders) | 2
Deep vein thrombosis (Vascular disorders) | 2
Dry mouth (Gastrointestinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Ear pain (Ear and labyrinth disorders) | 2
Faecal incontinence (Gastrointestinal disorders) | 2
Haematoma (Vascular disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Hypernatraemia (Metabolism and nutrition disorders) | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 2
Hypophagia (Metabolism and nutrition disorders) | 2
International normalised ratio increased (Investigations) | 2
Laceration (Injury, poisoning and procedural complications) | 2
Lymphocyte count decreased (Investigations) | 2
Malaise (General disorders) | 2
Migraine (Nervous system disorders) | 2
Mucosal inflammation (General disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Myoclonus (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 2
Peripheral swelling (General disorders) | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 2
Retching (Gastrointestinal disorders) | 2
Tachycardia (Cardiac disorders) | 2
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators have the right to publish and/or present study data after publication of the sponsor's multicenter study publication provided that the investigator shall (i) provide the sponsor a copy of any proposed publication or presentation generally thirty (30) days in advance of the submission; (ii) delete any confidential information of the sponsor; and (iii) delay submission for generally up to ninety (90) days to permit the sponsor to prepare and file intellectual property applications.

DOCUMENTS (2):
  • Study Protocol (2016-07-14): https://cdn.clinicaltrials.gov/large-docs/64/NCT02535364/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-09): https://cdn.clinicaltrials.gov/large-docs/64/NCT02535364/SAP_001.pdf